CLINICAL TRIAL: NCT07081191
Title: Dose-response Effect of Community Dance Programme on the Physical, Cognitive, Psychosocial Health of Pre-frail and Mildly Frail Older Adults: A Cluster Randomised Trial With Co-design Approach and Process Evaluation
Brief Title: Dose-response Effect of Community Dance Programme
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Vivien Xi WU, PhD, Assistant Professor Vivien Wu Xi, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NUS-IRB-2024-271; HCSAINV24jan-0003 (Other Grant/Funding Number: National Medical Research Council)
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Dance; Older Adults; Frailty at Older Adults; Active Ageing
Keywords: dance; Older adults; Frailty
MeSH Terms: conditions — Frailty | interventions — Cytidine Diphosphate

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The student dance instructors will be blinded to the allocation of the AACs to either the intervention or the active control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): 2 sessions per week of CDP (75 minutes per session) will be administered to the older adults at the various AACs over a period of 12 weeks. The face to face dance sessions will also be supported by dance instructional videos to help the seniors practice on their own time.
  Interventions: Behavioral: Dance
- Active control (Active Comparator): 1 session per week of CDP (60 minutes per session) will be administered to the older adults at the various AACs over a period of 12 weeks.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Dance — CDP was designed based on a 12-week dance curriculum, which involves 3 separate blocks of choreography of increasing complexity and intensity. According to World Health Organization, a minimum of 150 minutes of moderate intensity exercise would result in improvement in physical health, therefore, the intervention arm would involve 2 sessions of CDP, 75 minutes per session each week.
  Other Names: CDP
  Arms: Intervention arm
Behavioral: Active Control — CDP was designed based on a 12-week dance curriculum, which involves 3 separate blocks of choreography of increasing complexity and intensity. According to World Health Organization, a minimum of 150 minutes of moderate intensity exercise would result in improvement in physical health, therefore, the active control arm would only include 60 minutes of CDP (1 session) per week to assess the effect of CDP on the cognitive and physical health of older adults.
  Arms: Active control

SUMMARY:
The goal of this interventional study is to examine the dose-response effect of Community Dance Programme (CDP) on the physical, cognitive and psychological health of pre-frail and mildly frail community-dwelling older adults. The main questions it aims to answer are:

Hypothesis 1: Two sessions of CDP per week (75 minutes each) significantly increase the physical outcomes (i.e. CFS, EFS, SPPB, grip strength) of community-dwelling older adults as compared to one session of CDP per week.

Hypothesis 2: Two sessions of CDP per week significantly improve the cognitive outcomes (i.e. MoCA, SDMT) of community-dwelling older adults as compared to one session of CDP per week.

Hypothesis 3: Two sessions of CDP per week significantly improve the psychosocial outcomes (i.e. WHOQOL-OLD, De Jong Giervald Loneliness Scale, GPIC scale, SHS, SSQ) of community-dwelling older adults as compared to one session of CDP per week.

Intervention: The participants will be asked to attend two sessions of CDP per week for 12 weeks at their respective Active Ageing Centres (AACs).

Active control: The participants will be asked to attend one session of CDP per week for 12 weeks AACs.

* The participants will be asked to go to the AACs at baseline and after 12 weeks of CDP intervention for the collection of data.
* The participants will be asked to wear fitness trackers to track their heart rates during the CDP sessions to ensure that the dance curriculum is kept within the moderate intensity.

DETAILED DESCRIPTION:
Dance interventions have been shown beneficial for older adults, such as improving their physical health, cognitive function, as well as their psychosocial and emotional well-being by ameliorating depression, anxiety, and social isolation. A pilot study (NUS-IRB-2020-808) showed that those in the dancing group reported significantly higher quality of life (p=0.044). The qualitative findings provided insights that older adults enjoyed participating in the creatively crafted dance programme, while learning nature and world travel-based dance movements. Thus, this study aims to use data derived from the pilot study to design and conduct a definitive study to define the dose-response effect that a systematic dance programme may have on physical, cognitive, and psycho-social health in our local aging population.

A cluster-randomised trial with a co-design approach and process, evaluation will be applied. A qualitative approach with in-depth, face-to-face, focused group discussions (FGDs-needs assessment) will be conducted for stakeholders (older adults, AAC staff, and dance instructors) to understand their needs (e.g., factors promoting dance, measures to overcome common side effects of dance, social-cultural considerations) and seek their opinions further to develop the Community Dance Programme (CDP). CDP will be developed following the WHO ICOPE's guidelines and validated by a panel of multi-disciplinary experts. The participants will be randomly separated into 2 clusters: Intervention Clusters (2 sessions/week and 75 minutes/session) and Active Control Clusters (1 session/week and 1 hour/session). The interventional face to face sessions will be supported by instructional dance videos which allows the seniors to practice the dance on their own time.

12 weeks of dance sessions will be conducted. Objective assessments and self-reported questionnaires will be used pre and post-CDP. Outcome measures will include physical health (Short Physical Performance Battery, Edmonton Frailty Scale, biomarkers), cognitive function (Montreal Cognitive Assessment, Symbol Digit Modalities Test), psychosocial health (Geriatric Depression Scale, de Jong Gierveld Loneliness Scale, Subjective Happiness Scale, Social Support Questionnaire), and quality of life (WHOQOL).

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 to 85.
* Able to understand and communicate in either English or Mandarin.
* Able to give consent to participate.
* Able to commit for three months and able to achieve at least an attendance rate of 75% for the dance program.
* Lives within the community setting.
* Abbreviated Mental Test (AMT) score>= 8
* Obtain a score of less than or equal to 7 in Edmonton Frail Scale - Acute Care or less than or equal to 5 in Clinical Frailty Scale
* Able to ambulate with minimal assistance
* Willing to avoid other physical exercise during the interventional period.
* Consent to video and photography of the dance sessions and audio recording of the FGDs.

Exclusion Criteria:

* Abbreviated Mental Test (AMT) score of less than 8.
* A score of more than 7 on the Edmonton Frail Scale - Acute Care or a score of more than 5 on Clinical Frailty Scale
* Diagnosed with severe cognitive or psychiatric disorders.
* Have severe hearing or vision impairments
* Have medical conditions which results in limitation of dancing (e.g. walking aids, wheelchair etc.)
* Older adults with serious chronic diseases (e.g. postural hypotension etc.)
* Registered in any other dance group during the intervention period

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery | From enrollment to the end of the interventional period at 12 weeks.
  Evaluates the physical function. This instrument comprises physical tests of standing balance, gait speed, and chair stand. Each component (i.e., balance, gait speed, chair stand) will be scored from 0 to 4, with a score of 0 indicating inability to carry out the test and a score of 4 indicating perfect execution of the test. The total score ranges from 0 to 12, with higher scores indicating higher physical performance

SECONDARY OUTCOMES:
Clinical Frailty Scale | From enrollment to end of interventional period of 12 weeks
  This is a 9 point-scale which assesses the degree of frailty based on a visual chart which aids trained assessors to evaluate frailty. This scale depends on individual clinical judgement assess if the patient can independently perform tasks such as bathing, dressing, housework, going upstairs, going out alone, going shopping, taking care of finances, taking medications, and preparing meals. The higher the number, the more frail the individual. It is a tool that has been validated and widely used in local clinical and community settings.
Edmonton Frailty Scale - Acute Care | From enrollment to end of interventional period of 12 weeks
  This is an 11-item questionnaire that examines nine domains of frailty (i.e., cognition, general health status, functional independence, social support, medication use, nutrition, mood, continence, and functioning performance). The scores range from 0 to 17, with higher scores indicating higher levels of frailty. The scores can be categorized into five levels of frailty, namely: fit (0-3), vulnerable (4-5), mild frailty (6-7), Moderate frailty (8-9) and severe frailty (≥10).
  This instrument has been utilised and validated in a local tertiary hospital, with high acceptability and low inter-rater variability
Screening for Oral Frailty Tool | From enrollment to end of interventional period of 12 weeks
  The oral frailty scale comprises 6 items, including number of teeth, difficulty in swallowing, difficulty in chewing, difficulty in articulatory oral motor, dry mouth, and oral pain, and is assessed using a yes or no question. The correlations ranged from 0.40 to 0.66 when correlating each item with the total score of the scale. Using frailty and sarcopenia as criteria, the area under the curve for the SOFT was 0.71. The optimal cutoff for the SOFT was 2,
MOXY (muscle oxygenation) | From enrollment to the end of the interventional period of 12 weeks.
  MOXY (Moxy, Fortiori Design LLC, Minnesota, USA) is a non-invasive small wearable portable device that measures muscle oxygen saturation (SmO2), using near-infrared spectroscopy (NIRS) [38]. MOXY measures oxygen levels in the muscles of participants during exercise. Saliva sampling and MOXY oxygen monitoring are non-invasive procedures.
Examining the rate of DNA methylation | From enrollment to the end of the interventional period of 12 weeks
  DNA methylation analysis will be conducted on the saliva samples collected from the older adults to examine the DNA methylation patterns at specific DNA sites to detect epigenetic clocks that change with age.
Global Perception of Intergenerational Communications | From enrollment to the end of the interventional period of 12 weeks.
  The Revised Global Perceptions of Intergenerational Communication scale measures both inter and intra intergenerational communication based on four domains, namely: accommodation, non-accommodation, respect/obligation and avoidant communication. The revised GPIC scale has shown cronbach alpha score of 0.7 for the older participants for the respect-obligation factor and higher cronbach alpha scores of 0.79 and 0.77 for in group and out group respectively for the accommodation factor and 0.79 and 0.75 for the in-group and out-group respectively for the non-accommodation score. This indicates a high reliability for the tool.
Subjective Happiness Scale | From enrollment to the end of the interventional period of 12 weeks
  Using a "subjectivist" approach to the assessment of happiness, a 4-item measure of global subjective happiness was developed and validated in 14 studies with a total of 2732 participants. Results indicated that the Subjective Happiness Scale has high internal consistency, which was found to be stable across samples. Test-retest and self/peer correlations suggested good to excellent reliability, and construct validation studies of convergent and discriminant validity confirmed the use of this scale to measure the construct of subjective happiness
De Jong Gierveld Loneliness Scale | From enrollment to the end of the interventional period of 12 weeks
  Loneliness concerns the subjective evaluation of one's situation, characterised by either a smaller than desirable number of relationships with friends (social loneliness), or situations whereby the intimacy in confidant relationships one wishes for has not been realised (emotional loneliness) [44]. dJGLS-6 (six-item) will be used to measure social and emotional loneliness.
Social Support Questionnaire-6 | From enrollment to the end of the interventional period of 12 weeks
  This scale is developed by Sarason et al. [47]. It is used to measure the number of people providing support to an individual and the satisfaction level of the individual who received the support. The scale consists of 6 items. Rating of the items is from 1 (very dissatisfied) to 6 (very satisfied). With excellent Cronbach alphas of 0.90 and 0.93 for 2 respective domains, the scale has been proved to be valid and reliable.
WHOQOL-OLD | From enrollment to the end of the interventional period of 12 weeks
  WHOQOL-OLD for older adults to measure the quality of life for elderly. WHOQOL-OLD contain-ing six facets (including sensory abilities; autonomy; past, present, and future activities; social participation; death and dying; and intimacy), with four items in each facet [48]. Each of the facets has four items and therefore can obtain a possible score ranging from 4 to 20. The sum of the facet scores results in an overall QOL score.
Geriatric Depression Scale | From enrollment to the end of the interventional period of 12 weeks
  This scale contains 15 close-ended questions [42]. One point is allocated per question with the total scores below four indicating the absence of clinically depressive symptoms while scores between four and nine are indicative of mild to moderate depression. Scores of 10 or more are suggestive of a major depressive episode.

CONTACTS AND LOCATIONS:
Overall Officials: Vivien Wu Xi, Principal Investigator — National University of Singapore
Locations (1):
- Lion Befrienders' Active Ageing Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The data will be decoded and anonymised

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT07081191/Prot_SAP_000.pdf